CLINICAL TRIAL: NCT04689698
Title: Influence of Flossing Tape Therapy on the Range of Motion and Influencing of Fascial Chains in the Lower Limbs
Brief Title: The Effect of Flossing to Joint Range of Motion.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Malá Jitka, Clinical researcher, department of physiotherapy, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pisarčík, Flossing
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2020-12

CONDITIONS: Muscle, Ligament and Fascia Disorders
Keywords: Muscle chains, fascia, range of motion, viscosity.

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Diagnostic Test: Thomayer test

INTERVENTIONS:
Diagnostic Test: Thomayer test — Testing of the ankle in sagittal line and Thomayer test before and after flossing of sole.
  Other Names: Dorziflexion of an ankle

SUMMARY:
This research aims to verify the effect of therapy called "tissue flossing" on the range of motion and examine the impact of this treatment on the Superficial fascial backline, described by Myers. The research aims to verify whether the thick rubber bands used to create a certain degree of compression in a predetermined part of the musculoskeletal system can help to increase the range of motion (ROM) and whether this increase in motion can be achieved by influencing fascial chains even in distant parts of the musculoskeletal system, outside the primary therapeutic zone treated by the tissue flossing method. The research aims to verify and especially compare the patient's joints' range of motion before and immediately after the tissue flossing treatment. The results of the experiment clarify the influence of the tissue flossing therapy method on the range of motion at the application site, on the range of motion in other joints within the Superficial fascial backline described by Myers and last but not least to prove the existence of these fascial chains in the human body.

DETAILED DESCRIPTION:
Methodology:

The weight-bearing lunge test (WBLT) was used to evaluate the change in the ankle joint's range of motion. A simple forward bend test - the Thomayer test - was used to evaluate the therapy's effect on the Superficial fascial backline described by Myers. Both tests are non-invasive. Both tests can be used to evaluate the outcome of a given therapy objectively. Both tests are elementary to perform and highly standardized and commonly used in similar research.

After completing the entrance tests, the tissue flossing method is applied to each proband. The treatment alone does not typically last more than 20 minutes for any proband. As part of the tissue flossing treatment, both lower limbs of the proband will be treated. The "tissue flossing" method will be applied according to the authors' standard recommendations first to the plantar fascia area, then to the ankle joint. Finally, the last treated structure will be the area of fascia cruris. The duration of each application does not exceed 2 minutes. The order of individual applications is determined in advance as follows: right and then left plantar fascia, right and then left ankle joint and right and then left fascia cruris. Each application will be supplemented by the standard manual treatment or supplemented by the proband's active movement. After a total of 6 treatments, the therapeutic unit will be finished, and each proband will be re-examined using the same tests as before the treatment. If a given proband experiences any undesirable complications during the application of the "tissue flossing" method or applying the given method to the proband is subjectively unpleasant, the given treatment will be finished immediately.

ELIGIBILITY:
Inclusion Criteria:

* No previous experience with the tissue flossing method
* Each proband had to do recreational or elite sports

Exclusion Criteria:

* persons with an acute, especially infectious disease, person with an injury or persons in the process of recovery after an injury or illness
* vascular diseases

Ages: 19 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Measurement of range of motion of ankle in sagital line | 5 minutes
  Measurement without flossing of sole in natura
Measurement of range of motion of ankle in sagital line | 15 minutes
  Flossing of sole and than measurement after flossing of sole
Measurement of range of motion of lumbar spine in sagital line | 5 minutes
  Measurement before flossing of sole
Measurement of range of motion of lumbar spine in sagital line | 15 minutes
  Measurement after flossing of sole

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, PhDr.Ph.D., Principal Investigator — Charles University, Faculty of physical education and sport
Locations (1):
- Charles University, Prague, Czechia